CLINICAL TRIAL: NCT06580587
Title: A Clinical Study to Evaluate the Breast Milk, Plasma and Whole Blood Pharmacokinetics of MK-8527 in Healthy Lactating Female Participants
Brief Title: A Study of MK-8527 in Healthy Lactating Female Participants (MK-8527-009)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8527-009; MK-8527-009 (Other: MSD)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy; HIV Pre-exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-8527 (Experimental): Participants receive single oral dose of MK-8527 on Day 1
  Interventions: Drug: MK-8527

INTERVENTIONS:
Drug: MK-8527 — Oral administration

SUMMARY:
The goal of this study is to learn how MK-8527 moves through the healthy person's body over time. Researchers will measure for the amount of MK-8527 in breast milk that the baby will receive at many time points.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is at least 6 weeks postpartum at the time of administration of study intervention, following the delivery of a healthy singleton neonate
* Is willing and able to express breast milk at least twice daily for at least 120 hours after enrollment
* Is willing to discontinue breastfeeding from the time of administration of study intervention until at least 6 weeks following the administration of study intervention. This includes the avoidance of both directly breastfeeding and the administration of breast milk pumped during the above-specified time frame to the infant. Is willing to confirm with the site that the infant is able to bottle feed (breast milk) prior to Day 1 and that alternative nutrition (i.e., previously stored breast milk or infant formula) is available for feeding the infant through the 6-week post dose period

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, psychiatric, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Had mastitis within 30 days prior to administration of study drug
* Has a positive pregnancy test at the time of screening or prior to treatment allocation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy Lactating Female Participants
Enrollment: 12 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03-27 (Estimated); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to 120 hours (AUC0-120hrs) After Administration of a Single Oral Dose of MK-8527 in Breast Milk | Predose and at designated timepoints up to 120 hours postdose
  Breast milk samples will be collected to determine the AUC0-120hrs after administration of a single oral dose of MK-8527.
Maximum Breast Milk Concentration (Cmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 21 days postdose
  Breast milk samples will be collected to determine the Cmax after administration of a single oral dose of MK-8527.
Time to Maximum Breast Milk Concentration (Tmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 21 days postdose
  Breast milk samples will be collected to determine the Tmax after administration of a single oral dose of MK-8527.

SECONDARY OUTCOMES:
Mean Concentration of MK-8527 in Breast Milk After Administration of a Single Oral Dose | Predose and at designated timepoints up to 120 hours postdose
  Breast milk samples will be collected to determine the mean concentration of MK-8527.
Amount Excreted in Breast Milk From Time Zero to 120 Hours (Ae0-120hrs) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 120 hours postdose
  Breast milk samples will be collected to determine the Ae0-120hrs after administration of a single oral dose of MK-8527.
Area Under the Concentration-Time Curve from Time 0 to 120 hours (AUC0-120hrs) After Administration of a Single Oral Dose of MK-8527 in Blood | Predose and at designated timepoints up to 120 hours postdose
  Blood samples will be collected to determine AUC0-120hrs after administration of a single oral dose of MK-8527.
Area Under the Concentration-Time Curve from Time 0 to Time-Infinity (AUC0-Inf) After Administration of a Single Oral Dose of MK-8527 in Blood | Predose and at designated timepoints up to 21 days postdose
  Blood samples will be collected to determine AUC0-inf after administration of a single oral dose of MK-8527.
Maximum Blood Concentration (Cmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 21 days postdose
  Blood samples will be collected to determine the Cmax after administration of a single oral dose of MK-8527.
Time to Maximum Blood Concentration (Tmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 21 days postdose
  Blood samples will be collected to determine the Tmax after administration of a single oral dose of MK-8527.
Area Under the Concentration-Time Curve from Time 0 to 120hours (AUC0-120hrs) After Administration of a Single Oral Dose of MK-8527 in Plasma | Predose and at designated timepoints up to 120 hours postdose
  Plasma samples will be collected to determine AUC0-120hrs after administration of a single oral dose of MK-8527.
Area Under the Concentration-Time Curve from Time 0 to Time-Infinity (AUC0-Inf) After Administration of a Single Oral Dose of MK-8527 in Plasma | Predose and at designated timepoints up to 7 days postdose
  Plasma samples will be collected to determine AUC0-inf.
Maximum Plasma Concentration (Cmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 7 days postdose
  Plasma samples will be collected to determine the Cmax after administration of a single oral dose of MK-8527.
Time to Maximum Plasma Concentration (Tmax) After Administration of a Single Oral Dose of MK-8527 | Predose and at designated timepoints up to 7 days postdose
  Plasma samples will be collected to determine the Tmax after administration of a single oral dose of MK-8527.
Ratio of MK-8527 in Breast Milk to Blood After Administration of a Single Dose of MK-8527 | At designated timepoints up to 120 hours postdose
  Ratio of MK-8527 in breast milk to blood will be used to estimate dose of MK-8527.
Ratio of MK-8527 in Breast Milk to Plasma After Administration of a Single Oral Dose | At designated timepoints up to 120 hours postdose
  Ratio of MK-8527 in breast milk to plasma will be used to estimate dose of MK-8527.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO ( Site 0002), Springfield, Missouri
  - University of Pittsburgh Medical Center Magee-Womens Hospital ( Site 0001), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com